CLINICAL TRIAL: NCT00890136
Title: COpd and Domestic Endotoxin (CODE)
Brief Title: Chronic Obstructive Pulmonary Disease (COPD) and Domestic Endotoxin (CODE)
Acronym: CODE
Status: Completed | Type: Observational
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Environmental Health Sciences (NIEHS) (NIH)
Responsible Party: Sponsor
Other Study IDs: NA_00017777
Record Dates: First submitted 2009-04-27; First posted 2009-04-29 (Estimated); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease (COPD)
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood, sputum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This project aims to characterize the independent effect of domestic endotoxin exposure on health status, as well as pulmonary and systemic inflammation, in former smokers with COPD. Positive findings from this study would be clinically relevant, as they would provide evidence to support aggressive reduction of ongoing endotoxin exposure in patients with COPD. The investigators also hope to make a methodological advance in the field of endotoxin exposure assessment by elucidating whether settled dust and/or airborne endotoxin measurements are the more relevant exposure of interest in epidemiological studies of respiratory disease. To fulfill the specific aims, the investigators will conduct a longitudinal study, including 75 former smokers with COPD. All subjects will have indoor air monitoring, in-home settled dust collections, home inspections as well as assessments of health status, quality of life (QOL), lung function and pulmonary and systemic inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Patient reported physician diagnosis of COPD/Chronic Bronchitis/Emphysema
* Cigarette Smoking > 10 pack-years
* Age > 40 years
* Has not smoked > 1 year
* Post BD FEV1/FVC ≤ 70%
* Post BD FEV1 (% predicted) 30-80%
* Ability and willingness to provide consent

Exclusion Criteria:

* Non- English speaking
* Planning to move or live away from the home during the study period
* Co-morbid illnesses such as:

  * Current physician diagnosis of Asthma
  * Other pulmonary diseases
  * Systemic disease requiring treatment with immunosuppressive agents
  * Known alpha-1 antitrypsin deficiency
  * Occupational exposure with high endotoxin exposure
* Within the last 6 months Use of oral corticosteroids

Ages: 40 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Both Male and Female 40 years and older
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2008-07 (Actual); Primary Completion 2014-03 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
statistical analysis | one year

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Hansel, MD, MPH, Principal Investigator — Johns Hopkins University
Locations (1):
- Karina Romero, Baltimore, Maryland, United States